CLINICAL TRIAL: NCT01010061
Title: An Open-label, Multi-center, Three Arm Randomized Study to Investigate the Safety and Efficacy on Progression-free Survival of RO5072759 + Chlorambucil (GClb) Compared to Rituximab + Chlorambucil (RClb) or Chlorambucil (Clb) Alone in Previously Untreated CLL Patients With Comorbidities.
Brief Title: CLL11: A Study of Obinutuzumab (RO5072759 [GA101]) With Chlorambucil in Patients With Previously Untreated Chronic Lymphocytic Leukemia (Stage 1a)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: German CLL Study Group (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21004 (Stage 1a); 2009-012476-28; CLL11; NCT02035462 (obsolete NCT alias)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; Rituximab; Chlorambucil

ARMS (3):
- obinutuzumab + chlorambucil (GClb) (Experimental): Participants received 1000 mg obinutuzumab intravenous (IV) infusion, on Days 1 [first infusion split 100 mg on Day 1 and 900 mg on Day 2 as per protocol amendment], 8 and 15 in Cycle 1 and Day 1 in Cycles 2-6 (28-day cycles) plus chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle (6 Cycles).
  Interventions: Drug: obinutuzumab; Drug: chlorambucil
- rituximab + chlorambucil (RClb) (Active Comparator): Participants received 375 mg/m^2 rituximab IV infusion on Day 1 of Cycle 1 then 500 mg/m^2 IV infusions on Day 1 of Cycles 2-6 (28-day cycles) plus chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle (6 cycles).
  Interventions: Drug: rituximab; Drug: chlorambucil
- Chlorambucil (Clb) (Active Comparator): Participants received chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle (6 Cycles). Participants with Progressive Disease or within 6 months of follow-up were allowed to cross over to receive obinutuzumab + chlorambucil.
  Interventions: Drug: chlorambucil

INTERVENTIONS:
Drug: obinutuzumab — 1000 mg obinutuzumab intravenous (IV) infusion, on Days 1 [first infusion split 100 mg on Day 1 and 900 mg on Day 2 as per protocol amendment], 8 and 15 in Cycle 1 and Day 1 in Cycles 2-6 (28-day cycles).
  Other Names: RO5072759; GA101; GAZYVA®
  Arms: obinutuzumab + chlorambucil (GClb)
Drug: rituximab — 375 mg/m^2 rituximab intravenous (IV) infusion on Day 1 of Cycle 1 (Cycle duration is 28 days) then 500 mg/m^2 IV infusions on Day 1 of Cycles 2-6.
  Other Names: Rituxan®; MabThera®
  Arms: rituximab + chlorambucil (RClb)
Drug: chlorambucil — Chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle.

SUMMARY:
This open-label, randomized, 3-arm study will evaluate the efficacy and safety of obinutuzumab (RO5072759) in combination with chlorambucil as compared to rituximab plus chlorambucil or chlorambucil alone in patients with previously untreated chronic lymphocytic leukemia (CLL). Patients will be randomized 2:2:1 to receive a maximum of six 28-day cycles of either RO5072759 (1000 mg intravenous (iv) infusion, on days 1, 8 and 15 of cycle 1 and day 1 of cycles 2-6) plus chlorambucil (0.5 mg/kg orally, days 1 and 15 of cycles 1-6), or rituximab (iv infusion day 1, 375 mg/m^2 cycle 1, 500 mg/m^2 cycles 2-6) plus chlorambucil, or chlorambucil alone. Anticipated time on study treatment is >6 months and follow-up for disease-progression and safety will be at least 5 years. In the US, this trial is sponsored/managed by Genentech.

DETAILED DESCRIPTION:
Protocol BO21004 is divided into 3 separate Unique Protocol IDs for reporting results on clinicaltrials.gov because there are 3 separate primary analyses conducted at different time-points.

* BO21004 (Stage 1a) [NCT01010061] includes the analysis of 2 of the 3 arms obinutuzumab plus chlorambucil (Glb) compared to chlorambucil (Clb) reported here.
* BO21004 (Stage 1b) [NCT01998880] includes the analysis of 2 of the 3 arms rituximab plus chlorambucil (RClb) compared to chlorambucil (Clb) reported separately.
* BO21004 (Stage 2) [NCT02053610] includes the analysis of 2 of the 3 arms obinutuzumab plus chlorambucil (Glb) compared to rituximab plus chlorambucil (RClb) reported separately.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/=18 years
* Documented Cluster of Differentiation Antigen 20 (CD20) + B-Cell Chronic Lymphocytic Lymphoma (B-CLL)
* Previously untreated Chronic Lymphocytic Leukemia (CLL) requiring treatment according to the National Cancer Institute (NCI) criteria
* Total Cumulative Illness Rating Scale (CIRS) > 6 and/or creatinine clearance < 70 ml/min

Exclusion Criteria:

* Prior CLL therapy
* Transformation of CLL to aggressive Non-Hodgkin's Lymphoma (NHL) (Richter's transformation)
* History of other malignancy unless the malignancy has been in remission without treatment for >/=2 years prior to enrolment, and except for carcinoma in situ of the cervix, basal or squamous cell skin cancer, surgically treated low-grade prostate cancer, or ductal carcinoma in situ (DCIS) of the breast treated with lymphectomy alone
* Positive hepatitis serology (HBV, HCV) or positive HIV or Human T Cell Leukemia Virus (HTLV) testing
* Patients with active infection requiring systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (214):
- United States (5):
  - San Diego, California
  - Chicago, Illinois
  - Baltimore, Maryland
  - Green Bay, Wisconsin
  - Waukesha, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Rosario
- Australia (12):
  - Adelaide, New South Wales
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Liverpool, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Greenslopes, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Kurralta Park, South Australia
  - Frankston, Victoria
  - Melbourne, Victoria
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Brazil (5):
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São Paulo, São Paulo
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Vratsa
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Rimouski, Quebec
- Zagreb, Croatia
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Denmark (5):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Odense
  - Vejle
- Cairo, Egypt
- Estonia (2):
  - Tallinn
  - Tartu
- France (21):
  - Angers
  - Bobigny
  - Caen
  - Clermont-Ferrand
  - Créteil
  - Le Mans
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Reims
  - Rennes
  - Rouen
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (67):
  - Ahaus
  - Amberg
  - Ansbach
  - Bamberg
  - Berlin
  - Bonn
  - Bremen
  - Cologne
  - Delitzsch
  - Detmold
  - Dresden
  - Duisburg
  - Erlangen
  - Eschweiler
  - Essen
  - Esslingen am Neckar
  - Frankfurt
  - Frankfurt (Oder)
  - Frankfurt am Main
  - Frechen
  - Freiburg im Breisgau
  - Giessen
  - Göttingen
  - Greifswald
  - Hamburg
  - Hamm
  - Hanover
  - Heidelberg
  - Homburg/Saar
  - Kaiserslautern
  - Karlsruhe
  - Kempten
  - Kiel
  - Koblenz
  - Kronach
  - Landshut
  - Lebach
  - Leer
  - Lemgo
  - Loerrach
  - Lüdenscheid
  - Magedburg
  - Mainz
  - Mannheim
  - Mutlangen
  - München
  - Neunkirchen/Saar
  - Nuremberg
  - Oldenburg
  - Porta Westfalica
  - Ravensburg
  - Recklinghausen
  - Regensburg
  - Rostock
  - Rüsselsheim am Main
  - Saarbrücken
  - Sindelfingen
  - Stuttgart
  - Trier
  - Tübingen
  - Ulm
  - Villingen-Schwenningen
  - Weilheim
  - Wendlingen
  - Witten
  - Worms
  - Würzburg
- Hong Kong, Hong Kong
- Italy (11):
  - Cagliari
  - Cosenza
  - Ferrara
  - Genova
  - Messina
  - Milan
  - Modena
  - Orbassano
  - Roma
  - Terni
  - Torino
- Mexico (5):
  - Aguascalientes
  - Culiacán
  - Hermosillo
  - Monterrey
  - San Luis Potosí City
- Netherlands (4):
  - Delftzijl
  - Enschede
  - Leeuwarden
  - Nieuwegein
- New Zealand (2):
  - Auckland
  - Christchurch
- Romania (2):
  - Bucharest
  - Târgu Mureş
- Russia (6):
  - Kazan'
  - Nizhny Novgorod
  - Penza
  - Perm
  - Rostov-on-Don
  - Ufa
- Bratislava, Slovakia
- Spain (22):
  - Manresa, Barcelona
  - Sabadell, Barcelona
  - Jerez de la Frontera, Cadiz
  - Santander, Cantabria
  - Donostia / San Sebastian, Guipuzcoa
  - A Coruña, LA Coruña
  - Santiago de Compostela, LA Coruña
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - San Cristóbal de La Laguna, Tenerife
  - Gandia, Valencia
  - Barcelona
  - Jaén
  - Las Palmas
  - Madrid
  - Málaga
  - Murcia
  - Salamanca
  - Seville
  - Toledo
  - Valencia
  - Zaragoza
- Switzerland (7):
  - Aarau
  - Basel
  - Bern
  - Chur
  - Lucerne
  - Sankt Gallen
  - Zurich
- Thailand (2):
  - Bangkok
  - Khon Kaen
- United Kingdom (11):
  - Bournemouth
  - Cambridge
  - Canterbury
  - Cardiff
  - Cottingham
  - Edinburgh
  - Glasgow
  - Leicester
  - London
  - Nottingham
  - Sutton

REFERENCES:
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Jaramillo S, Agathangelidis A, Schneider C, Bahlo J, Robrecht S, Tausch E, Bloehdorn J, Hoechstetter M, Fischer K, Eichhorst B, Goede V, Hallek M, Dohner H, Rosenquist R, Ghia P, Stamatopoulos K, Stilgenbauer S. Prognostic impact of prevalent chronic lymphocytic leukemia stereotyped subsets: analysis within prospective clinical trials of the German CLL Study Group (GCLLSG). Haematologica. 2020 Nov 1;105(11):2598-2607. doi: 10.3324/haematol.2019.231027. PMID 33131249
- [Derived] Gibiansky E, Gibiansky L, Buchheit V, Frey N, Brewster M, Fingerle-Rowson G, Jamois C. Pharmacokinetics, exposure, efficacy and safety of obinutuzumab in rituximab-refractory follicular lymphoma patients in the GADOLIN phase III study. Br J Clin Pharmacol. 2019 Sep;85(9):1935-1945. doi: 10.1111/bcp.13974. Epub 2019 Jul 12. PMID 31050355
- [Derived] Goede V, Fischer K, Busch R, Engelke A, Eichhorst B, Wendtner CM, Chagorova T, de la Serna J, Dilhuydy MS, Illmer T, Opat S, Owen CJ, Samoylova O, Kreuzer KA, Stilgenbauer S, Dohner H, Langerak AW, Ritgen M, Kneba M, Asikanius E, Humphrey K, Wenger M, Hallek M. Obinutuzumab plus chlorambucil in patients with CLL and coexisting conditions. N Engl J Med. 2014 Mar 20;370(12):1101-10. doi: 10.1056/NEJMoa1313984. Epub 2014 Jan 8. PMID 24401022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 787 patients were enrolled in the study. Following a 6 patient safety run-in prior to randomization, 781 patients were randomized.
Pre-assignment Details: 589 patients were randomized to 1 of 3 treatment groups in 2:2:1 ratio: GClb (n=238), RClb (n=233) or Clb (n=118) in Stage 1 and an additional 192 randomized to GClb or RClb in Stage 2 [NCT02053610]. Stage 1 was divided for analysis into: Stage 1a (GClb vs Clb) n=356 reported here and Stage 1b (RClb vs Clb) [NCT01998880] reported separately.
Period: Overall Study
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Started | 238 | 118
Received Study Drug | 236 | 116
Completed | 190 (Completed=Completed treatment.) | 78
Not Completed | 48 | 40
Not completed — Adverse Events or Intercurrent Illness | 33 | 16
Not completed — Disease Progression | 2 | 8
Not completed — Withdrew Consent | 5 | 1
Not completed — Death | 3 | 6
Not completed — Administrative/Other | 0 | 1
Not completed — Refused Treatment/Did Not Cooperate | 2 | 0
Not completed — Insufficient Therapeutic Response | 1 | 5
Not completed — Violation of Selection Criteria | 0 | 1
Not completed — Did Not Receive Treatment | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the participants who were included in the Stage 1a analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb) | Total
Number analyzed (Participants) | 238 | 118 | 356
Age, Customized [Number; unit: participants]
  <65 years | 42 | 26 | 68
  >=65 years | 196 | 92 | 288
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 43 | 141
  Male | 140 | 75 | 215

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of progression, relapse, or death from any cause as assessed by the investigator. Progressive disease (PD) required at least one of the following: ≥50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, ≥50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, ≥50% increase in the enlargement of the liver and/or spleen, Transformation to a more aggressive histology or After treatment, the progression of any cytopenia (a decrease of hemoglobin levels >20 g/L or <10 g/dL or a decrease of platelet counts >50% or <100 x 10^9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L).
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Intent-to-treat population included all randomized participants. Patients without PFS events were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Months | 31.1 [26.5 to 35.6] | 11.1 [10.7 to 11.3]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified — Type I error controlled through closed test procedure; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.16 to 0.28] — Stratified by Binet stage at Baseline

2. Primary Outcome: Percentage of Participants With Progression Free Survival Events
Description: Percentage of Participants with Progression Free Survival Events: disease progression, relapse, or death.
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Percentage of participants | 72.7 | 90.7

3. Secondary Outcome: Progression Free Survival Based on Independent Review Committee (IRC) Data
Description: PFS was defined as the time from randomization to the first occurrence of progression, relapse, or death from any cause as assessed by Independent Review Committee. Progressive disease required at least one of the following: ≥50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, ≥50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, ≥50% increase in the enlargement of the liver and/or spleen, Transformation to a more aggressive histology or After treatment, the progression of any cytopenia (a decrease of hemoglobin levels >20 g/L or <10 g/dL or a decrease of platelet counts >50% or <100 x 10^9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L).
Time Frame: Randomization to clinical cutoff date of 9 May 2013 (median observation 22.8 months)
Population: Intent-to-treat population included all randomized participants. Patients without PFS events were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Months | 27.2 [23.5 to 33.0] | 11.2 [11.0 to 12.1]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.14 to 0.27] — Stratified by Binet stage at Baseline

4. Secondary Outcome: Percentage of Participants With Progression Free Survival Events Based on Independent Review Committee (IRC) Data
Description: Percentage of Participants with Progression Free Survival Events: progression, relapse, or death from any cause as assessed by an Independent Review Committee.
Time Frame: Randomization to clinical cutoff date of 9 May 2013 (median observation 22.8 months)
Population: Intent-to-treat population included all randomized participants. Participants without PFS events were censored.
Measure: Number; unit: Percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Percentage of participants | 37.4 | 76.3

5. Secondary Outcome: Percentage of Participants With End of Treatment Response (EOTR)
Description: EOTR was the first response assessment 56 days from the last dose according to the International Workshop on Chronic Lymphocytic Leukaemia (IWCLL) guidelines. CR required: Peripheral blood lymphocytes below 4 x 10^9/L, Absence of significant lymphadenopathy, No hepatomegaly, No splenomegaly, Absence of disease, Blood counts above the following values (Neutrophils >1.5 x 10^9/L, Platelets >100 x 10^9/L, Hemoglobin >11g/dL) and Bone marrow at least normocellular for age. CRi was CR with incomplete bone marrow recovery. PR required the following for at least 2 months from end of treatment: ≥50% decrease in peripheral blood lymphocyte count from the pre-treatment value AND Either a ≥ 50% reduction in lymphadenopathy OR ≥50% reduction of liver enlargement OR ≥50% reduction of spleen enlargement PLUS at least one of the following: Neutrophils >1.5 x 10^9/ or ≥50% increase, Platelets >100 x 10^9/L or ≥50% increase, Hemoglobin 11 g/dL or ≥50% increase.
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Participants from the Intent-to-treat population (all randomized participants) with data available for analysis. Participants who did not reach the 3 month Follow-up visit at the time of the clinical cutoff are excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Percentage of participants
  Complete Response (CR) | 17.2 [12.7 to 22.6] | 0.0 [0.0 to 3.1]
  Complete Response incomplete (CRi) | 4.2 [2 to 7.6] | 0.0 [0.0 to 3.1]
  Partial Response (PR) | 48.3 [41.8 to 54.9] | 28.8 [20.8 to 37.9]
  Nodular Partial Response (nPR) | 7.6 [4.5 to 11.7] | 2.5 [0.5 to 7.3]
  Stable Disease | 5 [2.6 to 8.6] | 22.9 [15.7 to 31.5]
  Progressive Disease | 4.2 [2.0 to 7.6] | 28.8 [20.8 to 37.9]
  No Response Assessment | 13.4 [NA to NA] — 95% CI not estimated. | 16.9 [NA to NA] — 95% CI not estimated.

6. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response according to IWCLL guidelines was defined as the percentage of patients with CR, CRi,PR or nPR. CR required all of the following: Peripheral blood lymphocytes below 4 x 10^9/L, Absence of significant lymphadenopathy, No hepatomegaly, No splenomegaly, Absence of disease, Blood counts above the following values (Neutrophils >1.5 x 10^9/L, Platelets >100 x 10^9/L, Hemoglobin >11g/dL) and Bone marrow at least normocellular for age. CRi was CR with incomplete bone marrow recovery. PR required the following for at least 2 months from end of treatment: ≥50% decrease in peripheral blood lymphocyte count from the pre-treatment value AND Either a ≥ 50% reduction in lymphadenopathy OR ≥50% reduction of liver enlargement OR ≥50% reduction of spleen enlargement PLUS at least one of the following: Neutrophils >1.5 x 10^9/ or ≥50% increase, Platelets >100 x 10^9/L or ≥50% increase, Hemoglobin 11 g/dL or ≥50% increase.
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Percentage of participants
  Complete Response (CR) | 26.5 [21.0 to 32.6] | 0.0 [0 to 3.1]
  Complete Response incomplete (CRi) | 2.5 [0.9 to 5.4] | 1.7 [0.2 to 6]
  Partial Response (PR) | 47.1 [40.6 to 53.6] | 31.4 [23.1 to 40.5]
  Nodular Partial Response (nPR) | 2.1 [0.7 to 4.8] | 0 [0 to 3.1]
  Stable Disease | 4.2 [2 to 7.6] | 21.2 [14.2 to 29.7]
  Progressive Disease | 4.2 [2.0 to 7.6] | 28.8 [20.8 to 37.9]
  No Response Assessment | 13.4 [NA to NA] — 95% CI was not estimated. | 16.9 [NA to NA] — 95% CI was not estimated.
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Includes subjects with best overall response: CR, CRi, PR or nPR; Test type: Superiority; p < 0.0001, Chi-squared; Difference in Response Rates = 45.1, 95% CI 2-sided [34.7 to 55.5]

7. Secondary Outcome: Event Free Survival
Description: Event-free survival (EFS) was defined as the time between date of randomization and the date of disease progression/relapse, death, or start of a new anti-leukemic therapy. Progressive disease as per IWCLL criteria required at least one of the following: ≥50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, ≥50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, ≥50% increase in the enlargement of the liver and/or spleen, Transformation to a more aggressive histology or After treatment, the progression of any cytopenia (a decrease of hemoglobin levels >20 g/L or <10 g/dL or a decrease of platelet counts >50% or <100 x 10^9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L).
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Intent-to-treat population included all randomized participants. Patients without EFS events were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Months | 28.7 [23.9 to 32.9] | 10.8 [8.0 to 11.1]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Test type: Superiority; p < 0.0001, Log Rank, Stratified; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.15 to 0.26] — Stratified by Binet stage at Baseline

8. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Intent-to-treat population included all randomized participants. Patients without OS events were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Months | NA [74.2 to NA] — The median survival time and upper limit of 95% CI could not be estimated due to a low number of deaths. | 66.7 [50.9 to NA] — The upper limit of 95% CI could not be estimated due to a low number of deaths.
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Test type: Superiority or Other; p = 0.0196, Log Rank, Stratified; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.49 to 0.94]

9. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the date the response [either Complete Response (CR) or Partial Response (PR)] was first recorded until the date of Disease Progression or death due to any cause. Response was assessed according IWCLL guidelines.
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Participants from the Intent-to-treat population (all randomized participants) with CR or PR. Participants without response were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 191 | 41
Months | 24.8 [22.1 to 33.5] | 5.1 [3.3 to 6.7]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (stratified) = 0.19, 95% CI 2-sided [0.13 to 0.28]

10. Secondary Outcome: Percentage of Participants With Molecular Remission at the End of Treatment
Description: Molecular remission was defined as a minimal residual disease (MRD)-negative result at the end of treatment (assessment that occurred between 56 days and 6 months of last treatment). Molecular remission was assessed for all patients using a blood sample. Additionally, a bone marrow sample was obtained from patients whom the investigator assumed to have a complete response, consistent with the IWCLL guidelines. A combined analysis of blood and bone marrow results was conducted. A patient was considered MRD negative if result was less than 1 chronic lymphocytic leukemia (CLL) cell in 10000 leukocytes (MRD value < 0.0001) based on the method of allele specific polymerase chain reaction (ASO-PCR).
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 166 | 90
Percentage of participants | 25 [18.9 to 32.6] | 0 [0.0 to 4.0]

11. Secondary Outcome: Time to Re-Treatment/New-antileukemic Therapy
Description: Time to re-treatment/new anti-leukemic therapy was defined as time between the date of randomization and the date of first intake of re-treatment or new anti-leukemic therapy.
Time Frame: Randomization to clinical cutoff date of 10 Oct 2017 (median observation 62.5 months from randomization)
Population: Intent-to-treat population included all randomized participants. Participants without events (re-treatment or new anti-leukemic therapy) were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
Months | 55.7 [47.4 to NA] — The upper level of the 95% CI was not reached. | 15.1 [11.7 to 18.0]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil (GClb) vs Chlorambucil (Clb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (stratified) = 0.25, 95% CI 2-sided [0.19 to 0.35]

12. Secondary Outcome: Pharmacokinetics of Obinutuzumab (RO5072759) in Combination With Chlorambucil (Clb)
Description: Blood samples were collected from all patients allocated to the GClb treatment arm pre- and post-dose Day 1 of Cycles 1 to 6 and were sent to a laboratory. The concentration of obinutzumab in serum was determined using a validated enzyme-linked immunosorbent assay (ELISA) and was reported in micrograms/milliliter (μg/mL).
Time Frame: Pre- and post-dose sampling on day 1 of cycles 1-6 (Up to 26.8 months)
Population: PK population includes all participants with PK data available at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 220
μg/mL
  Post-dose Cycle 1 (n=201) | 247 (41.6)
  Pre-dose Cycle 2 (n=198) | 227 (57.9)
  Post-dose Cycle 2 (n=197) | 587 (36.5)
  Pre-dose Cycle 3 (n=193) | 165 (68.7)
  Post-dose Cycle 3 (n=192) | 527 (39.7)
  Pre-dose Cycle 4 (n=191) | 156 (74.3)
  Post-dose Cycle 4 (n=189) | 535 (41.0)
  Pre-dose Cycle 5 (n=185) | 163 (72.4)
  Post-dose Cycle 5 (n=181) | 534 (39.1)
  Pre-dose Cycle 6 (n=185) | 181 (69.0)
  Post-dose Cycle 6 (n=183) | 525 (39.6)

13. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Questionnaire Score
Description: The EORTC Quality of Life Questionnaire QLQ-C30 was used to assess patient-reported outcomes (PRO) and symptom burden. The QLQ-C30 contains 30 items including the functional scales of physical functioning (5 items), role functioning (2 items), emotional functioning (4 items), cognitive functioning (2 items), social functioning (2 items) and symptom scales including fatigue (3 items), nausea and vomiting (2 items), and pain (4 items) and six single item scales on dyspnea, sleep disturbance, appetite loss, constipation, diarrhea and financial impact. Final scores are transformed such that they range from 0 - 100, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be of minimally important difference to participants. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Cycle 4 Day 1 (Cy4D1)
Population: ITT population. Here, n signifies the number of participants who were evaluated for specified categories.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
unit on a scale
  Appetite Loss Scale: Baseline (n=226, 111) | 18.1 (28.46) | 19.8 (29.26)
  Appetite Loss Scale: Cy4D1 (n=189, 92) | 10.2 (21.77) | 14.5 (24.36)
  Cognitive Functioning Scale: Baseline (n=227, 111) | 80.6 (21.35) | 81.8 (22.76)
  Cognitive Functioning Scale:Cy4D1 (n=190,93) | 83.9 (20.31) | 85.8 (18.54)
  Constipation Scale: Baseline (n=225, 111) | 14.8 (23.94) | 16.8 (26.92)
  Constipation Scale: Cy4D1 (n=188, 93) | 15.1 (25.16) | 12.5 (23.53)
  Diarrhoea Scale: Baseline (n=226, 110) | 9.3 (20.05) | 8.8 (18.98)
  Diarrhoea Scale: Cy4D1 (n=189, 93) | 9.3 (19.47) | 6.5 (14.95)
  Dyspnoea Scale: Baseline (n=225, 109) | 27.1 (29.89) | 23.9 (27.63)
  Dyspnoea: Cy4D1 (n=189, 91) | 15.9 (23.71) | 22.3 (26.78)
  Emotional Functioning Scale: Baseline (n=226, 111) | 73.8 (23.45) | 72.9 (25.7)
  Emotional Functioning Scale: Cy4D1(n=190,93) | 82.5 (18.62) | 80.6 (18.48)
  Fatigue Scale: Baseline (n=226, 111) | 38 (25.72) | 36.9 (27.01)
  Fatigue Scale: Cy4D1(n=189, 93) | 29.2 (20.39) | 30.8 (23.00)
  Financial Difficulties Scale: Baseline (n=224,110) | 8.9 (20.69) | 13.6 (25.26)
  Financial Difficulty Scale: Cy4D1(n=189,93) | 7.4 (17.64) | 9.3 (19.88)
  Nausea, Vomiting Scale: Baseline (n=227, 111) | 5 (11.18) | 7.4 (18.49)
  Nausea, Vomiting Scale: Cy4D1 (n=189,93) | 5.5 (11.51) | 7.5 (17.81)
  Pain scale: Baseline (n=228, 111) | 22.9 (27.57) | 21.5 (25.66)
  Pain scale: Cy4D1 (n=190, 93) | 17.9 (24.09) | 17.7 (25.98)
  Physical Functioning Scale: Baseline (n=228, 111) | 73.7 (19.86) | 77.3 (18.87)
  Physical Functioning Scale: Cy4D1(n=189,93) | 78.6 (18.71) | 80.9 (16.24)
  Global Health Status Scale: Baseline (n=226, 111) | 58.4 (22.8) | 57.4 (22.9)
  Global Health Status Scale: Cy4D1(n=189,93) | 66.7 (20.03) | 63.4 (20.56)
  Role Functioning Scale: Baseline(n=227,110) | 76.1 (26.18) | 74.7 (28.35)
  Role Functioning Scale: Cy4D1(n=189,93) | 79.7 (23.64) | 81.5 (21.35)
  Social Functioning Scale:Baseline(n=226,110) | 86.3 (22.52) | 83.3 (25.34)
  Social Functioning Scale: Cy4D1(n=190,93) | 87.8 (19.97) | 85.5 (19.38)
  Insomnia Scale: Baseline (n=228,111) | 29.4 (31.12) | 31.5 (32.98)
  Insomnia Scale: Cy4D1(n=189,93) | 20.6 (27.13) | 24.4 (29.13)

14. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) QLQ-CLL16 Questionnaire Score
Description: EORTC Quality of Life Questionnaire (QLQ-CLL16) module was used to assess patient-reported outcomes and symptom burden. The QLQ-CLL16 module includes three multi-item scales assessing fatigue (2 items), treatment side effects and disease symptoms (8 items), infection (4 items) and two single item scales on social activities and future health worries. Final scores are transformed such that they range from 0 - 100, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be of minimally important difference to participants. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Cycle 4 Day 1 (Cy4D1)
Population: ITT population. Here, n signifies the number of participants who were evaluated for specified categories.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb)
Number analyzed (Participants) | 238 | 118
unit on a scale
  Disease Effects Scale: Baseline (n=209, 102) | 23 (18.89) | 23.7 (20.18)
  Disease Effects Scale: Cy4D1 (n=176, 86) | 15.0 (15.12) | 15.9 (14.16)
  Fatigue Scale: Baseline (n=209, 102) | 31.2 (25.83) | 27.6 (24.65)
  Fatigue Scale: Cy4D1 (n=176, 86) | 20.9 (21.51) | 23.4 (22.20)
  Future Health: Baseline (n=206, 101) | 47.7 (32.14) | 50.8 (33.53)
  Future Health: Cy4D1 (n=175, 86) | 29.5 (31.74) | 39.1 (30.33)
  Infection Scale: Baseline (n=209, 102) | 12 (15.91) | 14.6 (17.97)
  Infection Scale: Cy4D1 (n=176, 86) | 8.9 (11.65) | 8.5 (10.70)
  Social Problems: Baseline (n=206, 100) | 24.3 (31.99) | 26.3 (33.26)
  Social Problems: Cy4D1 (n=175, 85) | 19.4 (27.75) | 22.0 (27.00)
  Treatment Side Effects Scale: Baseline (n=209,102) | 19.8 (17.7) | 17.2 (15.27)
  Treatment Side Effect Scale: Cy4D1(n=176,86) | 14.7 (14.68) | 15.6 (16.11)

ADVERSE EVENTS:
Time Frame: Randomization to clinical cutoff (median observation 42 months)
Description: Safety population included patients who received at least 1 dose of study drug. Adverse Events are reported for Stage 1a (GClb and Clb arms). In Stage 1a, 4 patients randomized to the RClb arm actually received obinutuzumab and were included in the GClb arm for analysis.
Groups:
- Crossover Subjects: Obinutuzumab + Chlorambucil (GClb): Subjects in Clb arm who progressed during/within 6 months after end of Clb treatment had opportunity to cross over to GClb arm at discretion of investigator. Subjects received 1000 mg obinutuzumab IV infusion, on Day 1 [First infusion split 100 mg on Day 1 and 900 mg on Day 2 as per protocol amendment], 8 and 15 in Cycle 1 and Day 1 of Cycles 2-6 (28-day cycles) plus chlorambucil 0.5 milligram per kilogram of body weight (mg/kg) orally on Day 1 and 15 of each 28-day cycle (6 Cycles).
Arm/Group | Obinutuzumab + Chlorambucil (GClb) | Chlorambucil (Clb) | Crossover Subjects: Obinutuzumab + Chlorambucil (GClb)
Serious Adverse Events (participants affected / at risk) | 113/241 | 45/116 | 8/30
Other Adverse Events (participants affected / at risk) | 215/241 | 89/116 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Chlorambucil (GClb) (N=241) | Chlorambucil (Clb) (N=116) | Crossover Subjects: Obinutuzumab + Chlorambucil (GClb) (N=30)
Pneumonia (Infections and infestations) | 10 | 4 | 1
Respiratory tract infection (Infections and infestations) | 2 | 3 | 0
Septic shock (Infections and infestations) | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 0 | 0
Sepsis (Infections and infestations) | 0 | 4 | 1
Infection (Infections and infestations) | 1 | 1 | 0
Liver abscess (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Stenotrophomonas sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 27 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 4 | 2 | 0
Cardiac failure (Cardiac disorders) | 3 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0
Diabetic macroangiopathy (Vascular disorders) | 1 | 0 | 0
Dry gangrene (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Fracture treatment (Surgical and medical procedures) | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Basosquamous Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Major depression (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Chlorambucil (GClb) (N=241) | Chlorambucil (Clb) (N=116) | Crossover Subjects: Obinutuzumab + Chlorambucil (GClb) (N=30)
Neutropenia (Blood and lymphatic system disorders) | 99 | 21 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 9 | 7
Anaemia (Blood and lymphatic system disorders) | 27 | 12 | 3
Leukopenia (Blood and lymphatic system disorders) | 17 | 0 | 5
Nausea (Gastrointestinal disorders) | 32 | 29 | 3
Diarrhoea (Gastrointestinal disorders) | 23 | 13 | 3
Constipation (Gastrointestinal disorders) | 17 | 12 | 2
Vomiting (Gastrointestinal disorders) | 13 | 14 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 147 | 0 | 15
Pyrexia (General disorders) | 25 | 8 | 2
Fatigue (General disorders) | 16 | 12 | 1
Asthenia (General disorders) | 17 | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 8 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 2
Bronchitis (Infections and infestations) | 10 | 8 | 1
Headache (Nervous system disorders) | 19 | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 9 | 2
Urinary tract infection (Infections and infestations) | 14 | 2 | 0
Viral Upper Respiratory Tract Infections (Infections and infestations) | 14 | 6 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.